CLINICAL TRIAL: NCT04733300
Title: Online Mindfulness-Based College for Young Adults (MBC)
Brief Title: Online Mindfulness-Based College for Young Adults
Acronym: MBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eric Loucks (Other)
Responsible Party: Sponsor-Investigator, Eric Loucks, Associate Professor, Brown University
Organization: Brown University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: #1608001570
Record Dates: First submitted 2020-10-21; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Depressive Symptoms; Loneliness; Sedentary Behavior; Mindfulness; Physical Activity; Diet; Sleep; Emotional Regulation; Alcohol Consumption, Youth; Stress, Psychological
Keywords: Emerging adult; Young Adult; Mindfulness; Randomized Controlled Trial
MeSH Terms: conditions — Depression; Sedentary Behavior; Motor Activity; Emotional Regulation; Underage Drinking; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The methodological approach includes a 3-arm trial of MBC (i.e, standard-dose vs. low-dose) vs. health education control, with n=100 per arm (total sample size 300 participants enrolled and randomized).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All study staff will be blinded to the participant treatment allocation to promote equipoise with the exception of the instructor and staff member coordinating participants within each course. Participants randomized to low vs standard dose MBC will not know which dose they received as all participants are requested to reserve 2.5 hours for the program each week. Participants however will be unmasked about if they received MBC vs. health education due to how different the programs are in content. Data analyses will be performed by a statistician blinded to treatment allocation type. The data manager will be able to break blinding if needed for safety. Circumstances for breaking the blind would be a large number of adverse experiences (>10% of enrolled participants reporting AEs rated as severe or life threatening) taking place in one or more study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based College - Standard Dose (Experimental): MBC standard dose is a 9-week, 9 session program providing systematic and intensive training in mindfulness meditation practices. The curriculum is grounded in the manualized and standardized Mindfulness-Based Stress Reduction (MBSR) curriculum. MBSR was adapted to the young adult life stage by: (1) Training mindfulness skills such as attention control, self-awareness and emotion regulation, using the MBSR curriculum, and (2) applying these skills to the health behaviors and priorities most relevant to young adults. Specific behaviors and priorities targeted are social relationships, sleep, stress, diet, physical activity, obesity, alcohol consumption, substance use, digital media use, and performance (e.g. athletic, artistic and academic). The intervention is administered live, online via a video conferencing platform. The standard dose class meets once a week for 2.5 hours for 9 weeks. There is also an all-day retreat that takes place around week 6 of the program.
  Interventions: Behavioral: Mindfulness-Based College for Young Adults
- Mindfulness-Based College - Low Dose (Experimental): The MBC low-dose program is mirrored after the standard MBC program (described previously); however, instead of meeting for 2.5 hours each week, the low-dose MBC program is abbreviated to meet for 1.5 hours each week for the 9 weeks. MBC low-dose will be administered live, online via the free video conferencing platform, Zoom.
  Interventions: Behavioral: Mindfulness-Based College for Young Adults
- Health education control group (Active Comparator): Those randomized to the health education control group will receive young adult-specific online health resources offered through www.youngwomenshealth.org and www.youngmenshealthsite.org. Both websites provide resources to improve mental and physical health, and include opportunities to ask health questions, and learn ways to improve mental and physical well-being.
  Interventions: Other: Health Education for Young Adults

INTERVENTIONS:
Behavioral: Mindfulness-Based College for Young Adults — MB-College (MBC) is a 9-week, 9 session curriculum providing systematic and intensive training in mindfulness meditation practices, applied to health behaviors relevant to young adults (18-29). The curriculum, which is based on the manualized and standardized Mindfulness-Based Stress Reduction (MBSR) curriculum is designed to teach participants how to integrate and apply mindfulness in their everyday lives to the range of challenges arising from medical and psychological conditions and life stresses.
  MBC will be administered live, online via a video conferencing platform to participants enrolled in the active arms of the study: (1) standard dose MBC and (2) low-dose MBC. Standard dose MBC meets once a week for 2.5 hours for 9 weeks, while low-dose MBC meets for 1.5 hours per week for 9 weeks. There is an all-day retreat that takes place around week six of the program that applies to both MBC programs.
  Other Names: Mindfulness-Based College standard dose; Mindfulness-Based College low-dose
  Arms: Mindfulness-Based College - Low Dose; Mindfulness-Based College - Standard Dose
Other: Health Education for Young Adults — The health education control group will receive young adult-specific online health resources offered through www.youngwomenshealth.org and www.youngmenshealthsite.org. Both websites provide resources to improve mental and physical health, and include opportunities to ask health questions, and learn ways to improve mental and physical well-being.
  Arms: Health education control group

SUMMARY:
MB-College (MBC) is an 9-week, 9 session program (i.e., the study intervention being tested in the RCT) providing systematic and intensive training in mindfulness meditation practices, applied to health behaviors relevant to college students and young adults.

The MBC intervention will be administered live, online via the free video conferencing platform, Zoom, to all eligible study participants enrolled in the active arms of the study. In addition to the 9-week, 9 session MBC class, referred to as "standard dose MBC" from here on out, investigators will also be testing a "low-dose MBC" version of the intervention, where each weekly session will run 1.5 hours in length rather than 2.5 hours.

This is a 3-arm randomized controlled trial. The standard-dose and low-dose versions of the MBC intervention will be compared to a third arm of the study, a health education active control group. Members of the control group will be offered the MBC class upon completion of the research study.

The Study Aims are to: (1) Evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). (2) Evaluate impacts of MBC standard-dose vs. MBC low-dose vs. health education control group on health conditions relevant for emerging adults, demonstrated to be influenced by MBC in a prior study, specifically depressive symptoms, loneliness, and sedentary activity. (3) Explore mechanisms by which MBC may exert effects on aforementioned health conditions, including interoceptive awareness, decentering, and perceived stress.

Participant Population: young adults aged 18-29 years of age, residing in the United States who screen eligible will be invited to enroll. Students will be screened using a two-part process taking place online. Research assessments at baseline and 3-month will take place digitally using Qualtrics, LLC (Provo, UT, USA) survey management tool. Participants will be sent secure links via email that can be accessed with their participant identification number.

Enrolled participants will be randomly assigned to one of three groups: (1) standard MBC; (2) low-dose MBC or (3) health education control group. The control group will be given the opportunity to participate in the intervention after the study MBC course is completed and follow-up assessments have been administered.

DETAILED DESCRIPTION:
Study Design The methodological approach includes a 3-arm trial of MB-College (i.e., standard-dose vs. low-dose) vs. enhanced usual care waitlist control, with n=100 per arm

All research assessments will take place digitally using Qualtrics, LLC (Provo, UT, USA) survey management tool. Participants will be sent secure links via email that can be accessed with their participant identification number. The MBC classes will be offered online via Zoom by a trained and certified MBC instructor.

Baseline assessment links will be sent to all enrolled participants and completed within four weeks of the start of the interventions. A single follow-up survey, "the three month follow up" will occur at least one day after and up to five weeks after the end of the intervention (i.e. the Week 8 class). Staff will prioritize having participants complete the surveys within the first three weeks of the assessment window, but will allow for participants to complete up to five weeks after. Additionally, the study will accept online survey completed outside the official follow up window if needed.

The total length of involvement for study participants will be around 3-4 months from the time of enrollment to the time of the final research assessment. The study interventions last 9 weeks and take place in the first two months for individuals in the standard-dose and low-dose intervention arms.

Participant Recruitment:

Participants will be recruited to participate in MBC primarily online using the following methods: (a) electronic distribution of the MBC advertisement cards via social media, such as Facebook, Twitter, Instagram, etc.; (b) emails sent to student listservs and through academic social networks;.(c) word of mouth through graduates of the MBC program and university staff interested in supporting the study; and (d) online information sessions offered by course instructor prior to the start of class.

Inclusion of women and minority groups - efforts will be made to recruit both women and minority students by intentionally advertising for the study in locations where said populations congregate/have a presence. Randomized groups will attempt to be balanced on gender, race-ethnicity, and level of education.

Screening Process Online Screening: Those who express interest in the study will complete an online screening assessment and availability form. Those who screen eligible based on the anonymous online screening (part 1 of 2) will be given the informed consent form online to read over and complete followed by an availability and contact form (part 2 of 2).

Informed Consent Informed consent will be administered and collected using digital forms through Qualtrics, LLC (Provo, UT, USA) from interested students who have screened eligible based on the anonymous online screener (part 1 or 2). The digital signature and informed consent document will be kept on file in a secure locations separate from participant data.

Randomization Process Participants will be randomly assigned to one of three groups: (1) the standard-dose MBC group; (2) the low-dose MBC group; or (3) the health education control group. A covariate adaptive randomization process will be used, balancing groups based on gender, race-ethnicity, and level of education.

Assessment Overview:

The following participant assessments will be administered to study participants:

1. Baseline Assessments -online baseline assessment will be completed within the four weeks leading up to the start of the online interventions.
2. 3-Month Follow Up Assessments - following the end of the nine-week interventions, participants will complete online follow up assessments similar to the assessments given at baseline.

Measures Descriptions:

1. Demographics: age, race/ethnicity, socioeconomic status, education, sexual orientation and gender orientation, student status, and employment.
2. Childhood socioeconomic status: retrospective reporting of parents' education, based on standardized questionnaires used in the Atherosclerosis Risk in Communities (ARIC) study.
3. Treatment expectancy: 6-item Credibility/ Expectancy questionnaire.
4. Depressive symptomatology: Assessed using Center for Epidemiologic Studies Depression Scale Revised (CESD-R). The CESD survey has been used extensively in the epidemiologic literature to assess depressive symptomatology. The scale was updated to the CESD-R by Van Dam et al., which allows diagnosable criteria similar to Diagnostic and Statistical Manual (DSM) of Mental Disorders.
5. Anxiety: Assessed using the validated Generalized Anxiety Disorder 7-item (GAD-7) scale.
6. Adverse Childhood Experiences: Measured using the standardized Childhood Trauma Questionnaire (CTQ) and the Childhood Experiences of Care and Abuse Inventory neglect subscale.
7. Medication use: Assessed directly from participants' medication bottles and self-report using standardized forms, including medication name, dose, frequency of use, and reason of use.
8. Substance use: questions taken from the National College Health Assessment II.
9. Alcohol consumption: additional self-report standardized questions assessing current alcohol consumption taken from the Behavioral Risk Factor Surveillance Survey (BRFSS).8
10. Physical Activity: Self-report physical activity is assessed using the International Physical Activity Questionnaire (IPAQ).
11. Fruit and Vegetable Consumption: self-report standardized questions assessing current fruit and vegetable consumption taken from Harvard Food Frequency Questionnaire modified to 3-items.
12. Sleep: Sleep quality and duration is assessed using the validated Pittsburgh Sleep Quality Index (PSQI).
13. Mindfulness: Assessed using the validated Five Facet Mindfulness Questionnaire Short Form 15-items.
14. Perceived stress: Assessed using the validated 14-item Perceived Stress Scale.
15. Interoceptive awareness: Assessed using the validated Multidimensional Assessment of Interoceptive Awareness (MAIA-2).
16. Loneliness: Assessed using the validated R-UCLA Loneliness Scale.
17. Global Health: individual physical, mental and social health are measured using the validated NIH PROMIS Global Health v1.2 scale and PROMIS-29+2.
18. Mindfulness attendance and practice questions will be administered to intervention group participants at the time of the 3 month follow up to get at mindfulness exposure and dose.
19. Ecological Momentary Assessment-Stress: assessed using 3-item scale developed by Creswell et al 2019.

Withdrawal during intervention Some amount of dropout during the study is anticipated, and therefore investigators may decide to over enroll in the waitlist group to account for this expected issue. If a participant in the intervention group decides to withdraw from the study during the MB-College course, they will be invited to still take part in the follow up assessments.

Confidentiality Randomly generated participant identification numbers will be assigned to students who consent to data collection. All questionnaires and tasks will be completed under the assigned participant identification numbers. Consent forms and personal identifiable information will be kept separate and securely away from participant identification numbers in a secure digital file on closed network servers.

Blinding All study staff will be blinded to the participant treatment allocation with the exception of the instructor and staff member coordinating participants within each course. All staff monitoring participant assessments and survey completion will be blinded to the participant treatment allocation to promote equipoise. Data analyses will be performed by a statistician blinded to treatment allocation type. The data manager will be able to break blinding if needed for safety. Circumstances for breaking the blind would be a large number of adverse experiences (>10% of enrolled participants reporting AEs rated as severe or life threatening) taking place in one or more study group.

Acceptability Assessed via acceptability ratings using the validated Client Satisfaction Questionnaire (Cronbach's alpha=0.93), class attendance rates (proportion of eligible participants who complete MB-College, missing no more than 3 classes) and the Net Promoter Score.

Feasibility Assessed via (a) participant recruitment rates, (b) participant retention rates, and (c) treatment fidelity assessments, via delivery of treatment per protocol (assessed via percent adherence of instructors to curriculum guide module), receipt of treatment (assessed by class attendance), and enactment of treatment skills (assessed by home practice completion, mindfulness levels).

Ecological Momentary Assessments:

A 3-item customized measure of stress will be administered using time contingent ecological momentary assessments. SMS will be administered using Qualtrics SMS service sent to participants' personal phones. The numbers will be loaded into Qualtrics de-identified using participant ID numbers. The SMS messaging will be 1 way with participants completing the survey through a mobile link. The survey will be sent at baseline and follow-up assessments every day for 1 week 4 times per day between 10:00 am and 11:00 pm. The survey as well as assessment schedule were tested in a randomized controlled trials (n=153) and the researchers who conducted the study advised on the implementation for this pilot study.

Fidelity Monitoring:

Intervention fidelity will be ensured by (1) rigorous, program specific training for the instructor with feedback, (2) recording of all sessions with a 10% quality audit reviewed with instructor after each cohort, (3) monitoring participant attendance, home practice of treatment skills, and understanding of skills, and (4) a comprehensive mixed methods approach (e.g. daily practice logs) for understanding of treatment enactment.

Follow-up visits Follow-up surveys will be digitally distributed and completed within the pre-defined assessment windows previously outlined. Questionnaires and assessments administered at 3-months follow-up are identical to those administered at baseline with the exception that questionnaires for which the answers should not change or be informative (age, race/ethnicity, education, childhood socioeconomic status) are not given at follow-ups. In addition, adverse events are monitored and documented at each of the follow-up periods as well as throughout the duration of an individual's study involvement.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years of age
* Able to read, write, and speak in English
* Access to a computer, tablet, or smart phone device in order to complete online assessments and participate in the online interventions
* Reside in the United States during the research study

Exclusion Criteria:

* Current, regular mindfulness meditation practice ≥1 time per week
* Untreated, pre-existing mental health conditions, including borderline disorder, schizophrenia or psychosis, obsessive-compulsive disorder, panic attacks, alcohol or substance abuse, and eating disorders, who are not in regular care of a clinician. These participants are excluded as they may require additional or specialized treatment not able to be provided by the study or are already participating in practices similar to the intervention.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of online MBC as measured by participation rates | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Feasibility will be assessed via three measures. One measure of feasibility will be participant recruitment rates. See other primary outcomes for other measures used.
Feasibility of online MBC as measured by retention rates | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Feasibility will be assessed via three measures. One measure of feasibility will be participant retention rates. See other primary outcomes for other measures used.
Feasibility of online MBC as measured by treatment fidelity: Treatment per protocol | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Feasibility will be assessed via three measures. One measure of feasibility will be treatment fidelity (i.e., treatment per protocol), which will be assessed via the percent adherence of instructors to the MBC curriculum guide.
Feasibility of online MBC as measured by treatment fidelity: Receipt of treatment | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Feasibility will be assessed via three measures. One measure of feasibility will be treatment fidelity (i.e., receipt of treatment), which will be assessed by class attendance.
Feasibility of online MBC as measured by treatment fidelity: Enactment of treatment skills | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Feasibility will be assessed via three measures. One measure of feasibility will be treatment fidelity (i.e., enactment of treatment skills), which will be assessed by home practice completion.
Acceptability of online MBC as measured by the Client Satisfaction Questionnaire | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Acceptability will be assessed using three measures. One such measure of acceptability will be via acceptability ratings using the validated 8-item Client Satisfaction Questionnaire (CSQ-8). Scores for the CSQ-8 range from 8 to 32, with higher values indicating higher satisfaction. See other primary outcomes for other measures used.
Acceptability of online MBC as measured by class attendance | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Acceptability will be assessed using three measures. One such measure of acceptability will be class attendance rates (i.e., proportion of eligible participants who complete MBC, missing no more than 3 classes). See other primary outcomes for other measures used.
Acceptability of online MBC as measured by the Net Promoter Score | 3 months
  The primary aim of the study is to evaluate feasibility and acceptability of MBC delivered in two online formats (standard dose vs. low dose). Acceptability will be assessed using three measures. One such measure of acceptability will be via the Net Promoter Score (NPS). NPS scores range from 0 to 10, with higher values indicating higher ratings. The overall NPS for the program is determined by taking the percentage of participants who promoted the program (NPS of 9 or 10) and subtracting the percentage of participants who gave a score of 6 or lower. Neutral scores of 7 and 8 are not included in the calculation of overall NPS. See other primary outcomes for other measures used.

SECONDARY OUTCOMES:
Impact of online MBC on depressive symptoms | 3 months
  Evaluate impacts of MBC standard-dose vs. MBC low-dose vs. the health education active control on health conditions relevant for emerging adults, demonstrated to be influenced by MBC in a prior study, specifically depressive symptoms, loneliness, and sedentary activity. Depressive symptomatology will be assessed using Center for Epidemiologic Studies Depression Scale Revised (CESD-R). The CESD survey has been used extensively in the epidemiologic literature to assess depressive symptomatology. The scale was updated to the CESD-R by Van Dam et al., which allows diagnosable criteria similar to Diagnostic and Statistical Manual (DSM) of Mental Disorders. Total scores to the CESD-R scale range from 0 to 60, with higher values indicating greater depressive symptomology.
Impact of online MBC on loneliness | 3 months
  Evaluate impacts of MBC standard-dose vs. MBC low-dose vs. the health education active control on health conditions relevant for emerging adults, demonstrated to be influenced by MBC in a prior study, specifically depressive symptoms, loneliness, and sedentary activity. Loneliness will be assessed using the validated R-UCLA Loneliness Scale. Scores range from 20 to 80 with higher scores indicating greater levels of loneliness.
Impact of online MBC on sedentary activity | 3 months
  Evaluate impacts of MBC standard-dose vs. MBC low-dose vs. the health education active control on health conditions relevant for emerging adults, demonstrated to be influenced by MBC in a prior study, specifically depressive symptoms, loneliness, and sedentary activity. Sedentary activity will be assessed using the International Physical Activity Questionnaire (IPAQ). The IPAQ allows for two forms of scoring. Results can be reported in categories (e.g., low activity levels, moderate activity levels, or high activity levels with cutoff points being set by current health standards) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Explore mechanisms (i.e., interoceptive awareness) by which online MBC may influence health outcomes | 3 months
  Explore mechanisms by which MBC may exert effects on aforementioned health conditions. Interoceptive awareness will be assessed using the validated Multidimensional Assessment of Interoceptive Awareness (MAIA-2). The MAIA-2 reports average scores for eight distinct subscales (i.e., noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting). The mean scores calculated can range from 0 to 5 with higher scores indicating greater levels of interoceptive awareness. An overall mean score of the subscales will be the primary outcome.
Explore mechanisms (i.e., decentering) by which online MBC may influence health outcomes | 3 months
  Explore mechanisms by which MBC may exert effects on aforementioned health conditions. Decentering will be assessed using the validated Experiences Questionnaire (EQ). Scores range from 11 to 55 with higher scores indicating greater levels of decentering, thought to be a positive attribute.
Explore mechanisms (i.e., perceived stress) by which online MBC may influence health outcomes | 3 months
  Explore mechanisms by which MBC may exert effects on aforementioned health conditions. Perceived stress will be measured using the validated 14-item Perceived Stress Scale (PSS-14). Scores range from 0 to 56 with higher scores indicating greater perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Loucks, PhD, Principal Investigator — Mindfulness Center at Brown University
Locations (1):
- Mindfulness Center at Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
External researchers interested in utilizing these data will be encouraged to do so provided they adhere to participant confidentiality requirements stipulated by the research study protection of human subjects protocol and the Brown University IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1.5 years of study completion.
Access Criteria: Please contact the principal investigator, Eric Loucks, at eric.loucks@brown.edu.